CLINICAL TRIAL: NCT04764539
Title: Video Assisted Speech Technology to Enhance Functional Language Abilities in Individuals With Autism Spectrum Disorder
Brief Title: Video Assisted Speech Technology to Enhance Motor Planning for Speech
Acronym: VAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iTherapy, LLC (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Lois Brady, Principal Investigator, iTherapy, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R43DC018447-01 (NIH); 1R43DC018447-01 (NIH)
Record Dates: First submitted 2021-02-09; First posted 2021-02-21 (Actual); Results first posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Autism Spectrum Disorder; Apraxia of Speech
Keywords: autism; apraxia; speech therapy; speech pathology; nonverbal
MeSH Terms: conditions — Autism Spectrum Disorder; Apraxias; Autistic Disorder; Communication Disorders

STUDY DESIGN:
Intervention Model Description: Six children with ASD, between the ages of 4 and 8, were recruited to participate in a 12-sessions-long study that utilized the Video-Assisted Speech Therapy (VAST) application. The participants were divided into two groups: one which received the VR-integrated prototype, and one that received a 2D application on a tablet. Each session was approximately 15 minutes long (+/- 5 minutes), occurring twice per week.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stimuli administered via 2D format on an iPad Pro (Active Comparator): Participants were given the Video-Assisted Speech Therapy (VAST) video-modeling stimuli in a 2D format (iPad Pro). Three children with ASD, between the ages of 4 and 8, participated in a 14-sessions-long study that utilized the tablet-based VAST application. Sessions were held twice a week with each lasting approximately 15 minutes (i.e. +/- 5 minutes).
  Interventions: Behavioral: Video Assisted Speech Therapy (VAST)
- Stimuli administered in 3D format via VR goggles and bone conduction headphones (Active Comparator): Participants were given the Video-Assisted Speech Therapy (VAST) video-modeling stimuli in a VR format paired with a custom 3D-printed VR headset. Three children with ASD, between the ages of 4 and 8, participated in a 14-sessions-long study that utilized a 3D VR-integrated VAST prototype with bone conduction audio. Sessions were held twice a week with each lasting approximately 15 min (i.e. +/- 5 minutes).
  Interventions: Behavioral: Video Assisted Speech Therapy (VAST)

INTERVENTIONS:
Behavioral: Video Assisted Speech Therapy (VAST) — Six children with ASD, between the ages of 4 and 8, participated in a 14-sessions-long study that utilized the VR-integrated and the tablet-based VAST application. Three subjects received a 3D VR-integrated, bone conduction VAST prototype, while the remaining group of three received a tablet with a 2D version of the software. Sessions were held twice a week with each lasting approximately 15 minutes (i.e. +/- 5 minutes).

SUMMARY:
Nearly 3.5 million Americans are diagnosed with Autistic Spectrum Disorder (ASD), a communication disorder that causes skill limitations in the areas of language acquisition, sensory integration, and behavior. This lack of functional language ability limits conversation to its most basic parts, making daily tasks difficult for minimally to non-verbal individuals to achieve. iTherapy is developing the VAST platform, a personalized educational experience for students with ASD by creating a virtual reality-based video-modeling program to stimulate engagement and speech production practice, ultimately providing those with ASD an opportunity to enhance their quality of life by increasing their speech abilities which will enable them to build social networks and handle the events of daily life.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental communication disorder resulting in functional language and behavioral delays affecting over 3.5 million Americans. These delays vary with the severity of symptoms that present in ASD but often result in limited speech and increased communication challenges. Alongside linguistic acquisition, oral motor coordination is a crucial part of speech production.

Current clinical techniques have shown varying degrees of efficacy in improving functional language proficiency. Most techniques follow a drill-like procedure, where the child is made to repeat various sounds and phrases until they are retained. However, such a process requires potentially over twenty therapy sessions to show improvement which may then only be focused on one aspect of speech. This significantly limits the linguistic and social skills a student will acquire. To improve the efficacy of these therapy sessions, new technology must be developed to provide the most effective educational experience.

Video-assisted speech technology (VAST) is a method of using a video of a close-up model of the mouth and speaking simultaneously with it. Rather than present the individual with a static photograph of the initial phoneme, the entire sequence of oral movements can be presented sequentially via video-recorded segments of the orofacial area producing connected speech, combining best practices, video modeling, and literacy with auditory cues to provide unprecedented support the development of vocabulary, word combinations and communication.

In this SBIR Phase I proposal, iTherapy will develop a personalized educational experience for students with ASD by creating a virtual reality (VR) based VAST program to stimulate engagement and speech production practice. VR offers several benefits as a therapy technique: overcoming sensory difficulties, more effectively generalizing information, employing visual learning, and providing individualized treatment. As a user moves through the stages of the program, they will be immersed in a proactive environment where they will engross themselves with continuous content.

Rather than present the individual with a static photograph of the initial phoneme, the entire sequence of oral movements can be presented sequentially via VR-modelled segments of the orofacial area producing connected speech, combining best practices, video modeling, music therapy, and literacy with auditory cues to provide unprecedented support the development of vocabulary, word combinations and communication. The innovation will be a video series of a realistic VR mouth which will require the use of an app on a tablet or a smartphone, VR goggles, and bone conduction headphones.

ELIGIBILITY:
Inclusion Criteria:

* Nonverbal-minimally verbal children (0-5 words)
* Diagnosis of Autism Spectrum Disorder

Exclusion Criteria:

* No history of seizures for participating with VR goggles.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- All research was conducted via tele-research due to COVID-19, Vallejo, California, United States

IPD SHARING:
Plan to Share IPD: No
All data from individual participants will be kept private.

REFERENCES:
- [Background] Baio J, Wiggins L, Christensen DL, Maenner MJ, Daniels J, Warren Z, Kurzius-Spencer M, Zahorodny W, Robinson Rosenberg C, White T, Durkin MS, Imm P, Nikolaou L, Yeargin-Allsopp M, Lee LC, Harrington R, Lopez M, Fitzgerald RT, Hewitt A, Pettygrove S, Constantino JN, Vehorn A, Shenouda J, Hall-Lande J, Van Naarden Braun K, Dowling NF. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2014. MMWR Surveill Summ. 2018 Apr 27;67(6):1-23. doi: 10.15585/mmwr.ss6706a1. PMID 29701730
- [Background] Autism Spectrum Disorder: Communication Problems in Children. (2018, August 30). Retrieved from https://www.nidcd.nih.gov/health/autism-spectrum-disorder-communication-problems-children
- [Background] Maas E, Robin DA, Austermann Hula SN, Freedman SE, Wulf G, Ballard KJ, Schmidt RA. Principles of motor learning in treatment of motor speech disorders. Am J Speech Lang Pathol. 2008 Aug;17(3):277-98. doi: 10.1044/1058-0360(2008/025). PMID 18663111
- [Background] Bent S, Hendren RL. Complementary and alternative treatments for autism part 1: evidence-supported treatments. AMA J Ethics. 2015 Apr 1;17(4):369-74. doi: 10.1001/journalofethics.2015.17.4.sect1-1504. No abstract available. PMID 25901707
- [Background] Lord, C., & Paul, R. (1997). Language and communication in autism. In D. Cohen & F. Volkmar (Eds.), Handbook of autism and pervasive developmental disorders (pp. 195-225). New York, NY: Wiley.
- [Background] Jang J, Matson JL, Williams LW, Tureck K, Goldin RL, Cervantes PE. RETRACTED: Rates of comorbid symptoms in children with ASD, ADHD, and comorbid ASD and ADHD. Res Dev Disabil. 2013 Aug;34(8):2369-78. doi: 10.1016/j.ridd.2013.04.021. Epub 2013 May 22. PMID 23708709
- [Background] Battle DE. Diagnostic and Statistical Manual of Mental Disorders (DSM). Codas. 2013;25(2):191-2. doi: 10.1590/s2317-17822013000200017. No abstract available. PMID 24413388
- [Background] Symptoms and Diagnosis of ADHD | CDC. (n.d.). Retrieved from https://www.cdc.gov/ncbddd/adhd/diagnosis.html.
- [Background] Sarah Parsons & Sue Cobb (2011) State-of-the-art of virtual reality technologies for children on the autism spectrum, European Journal of Special Needs Education, 26:3, 355-366, DOI: 10.1080/08856257.2011.593831
- [Background] Strickland DC, McAllister D, Coles CD, Osborne S. An Evolution of Virtual Reality Training Designs for Children With Autism and Fetal Alcohol Spectrum Disorders. Top Lang Disord. 2007 Jul 1;27(3):226-241. doi: 10.1097/01.tld.0000285357.95426.72. PMID 20072702
- [Background] Evers, K., Noens, I., Steyaert, J., & Wagemans, J. (2011). Combining strengths and weaknesses in visual perception of children with an autism spectrum disorder: Perceptual matching of facial expressions. Research in Autism Spectrum Disorders,5(4), 1327-1342. doi:10.1016/j.rasd.2011.01.004
- [Background] Strickland D, Marcus LM, Mesibov GB, Hogan K. Brief report: two case studies using virtual reality as a learning tool for autistic children. J Autism Dev Disord. 1996 Dec;26(6):651-9. doi: 10.1007/BF02172354. PMID 8986851
- [Background] Handbook of Sensory Physiology - rd.springer.com. (n.d.). Retrieved from https://rd.springer.com/content/pdf/bfm:978-3-642-88658-4/1.pdf
- [Background] Why Speech Rate? Why are results inconclusive? (n.d.). Retrieved from https://www.asha.org/Events/convention/handouts/2007/1337_Chon_Hee_Cheong/ Brown, R. (1973) A First Language London: Allen and Unwin.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Stimuli Administered Via 2D Format on an iPad Pro: Three children with ASD, between the ages of 4 and 8, participated in a 14-sessions-long study that utilized the tablet-based Video-Assisted Speech Therapy (VAST) application. Sessions were held twice a week with each lasting approximately 15 minutes (i.e. +/- 5 minutes).
- Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones: Three children with ASD, between the ages of 4 and 8, participated in a 14-sessions-long study that utilized a 3D VR-integrated Video-Assisted Speech Therapy (VAST) application, which paired bone conduction audio within a 3D-printed headset prototype. Sessions were held twice a week with each lasting approximately 15 minutes (i.e. +/- 5 minutes).
- Total: Total of all reporting groups
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 3 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.75 (2.113) | 6 (1.938) | 5.875 (1.818)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Length of Utterance (MLU)
Description: Participants (aged 4 to 8 years) were given a pre- and post-test 15-minute language sample. MLU was calculated for tests and gain from pre-test to post-test was compared.
  NOTE: This measure is calculated based on a change in the number of morphemes per utterance during pre-test and post-test language samples. During a five-minute period, two licensed speech-language pathologists (SLP) observed a parent interacting and talking with their child. Parents Both SLPs transcribed the subjects' speech and calculated a mean length of utterance (MLU) for each subject. MLU was calculated by determining how many bound and free morphemes were included within every spoken utterance produced by a subject. The total number of morphemes produced within the 5-minute period were then divided by total number of utterances, which then produced the MLU for each subject. This procedure was use for determining MLU in both the pre- and post-testing procedures.
Time Frame: Seven weeks--each subject participated in the study twice a week over a 7-week period for a total of 14 sessions. The first and last sessions (session #1 and session #14) were reserved for pre-test and post-test language sample collection and assessment.
Population: All participants for each respective group.
Measure: Mean (Standard Deviation); unit: Morphemes per utterance
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
Number analyzed (Participants) | 3 | 3
Morphemes per utterance | 0.5387 (0.4119) | 0.2987 (0.4977)
Statistical Analysis 1: Comparison: Stimuli Administered Via 2D Format on an iPad Pro vs Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; The Mean Length of Utterance (MLU) will not increase from baseline for the either the iPad Pro or VR goggle participant group after having used the VAST system for 2 months; Test type: Superiority; p < 0.555, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.276 to 0.796], Standard Deviation 0.294 — Difference = (VR goggles group - iPad Pro group)
Statistical Analysis 2: Comparison: Stimuli Administered Via 2D Format on an iPad Pro; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.2128, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 0.5383, 95% CI 2-sided [-0.471 to 1.548], Standard Deviation 0.659 — Difference = (iPad Pro group Post-Treatment - iPad Pro group Pre-Treatment)
Statistical Analysis 3: Comparison: Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.533, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 0.298, 95% CI 2-sided [-0.915 to 1.511], Standard Deviation 0.365 — Difference = (VR goggles group Post-Treatment - VR goggles group Pre-Treatment)

2. Primary Outcome: Change in Percentage of Correctly Transcribed Words Using Automatic Speech Recognition
Description: 15-minute pre- and post-testing was performed using speech recognition software and transcribed by a licensed speech pathologist. Differences pre and post intervention were compared across group and within groups.
  NOTE: During our assessment, we used Google's native closed captioning function (a tool which uses machine learning to recognize and transcribe speech) and a third party app, Tactiq Pins, which allows users to keep a transcript of all speaker utterances during a call. We compared our video to the Tactiq Pin transcripts in order to measure any change in the amount of accurately transcribed spoken words between pre-test and post-test language samples. Specific transcription results for each group can be found in the data tables provided.
Time Frame: as for outcome 1
Population: All participants for each respective group.
Measure: Mean (Standard Deviation); unit: % of correctly transcribed words
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
Number analyzed (Participants) | 3 | 3
% of correctly transcribed words | 1.388 (1.966) | 0 (0)
Statistical Analysis 1: Comparison: Stimuli Administered Via 2D Format on an iPad Pro vs Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; The percentage of correctly transcribed words using automatic speech recognition will not increase from baseline for the either the iPad Pro or VR goggle participant group after having used the VAST system for 2 months; Test type: Superiority; p < 0.289, ANOVA — Sample size too small for statistical power. In addition, automated speech recognition for child speech had a very poor state-of-the-art at the time of this study; Mean Difference (Final Values) = 1.388, 95% CI 2-sided [-1.763 to 4.539], Standard Deviation 1.7 — Difference = (iPad Pro group - VR goggles group)

3. Primary Outcome: Change in Articulation Accuracy
Description: Change in % of correct phonemes in each attempted stimulus
Time Frame: as for outcome 1
Population: All participants for each respective group.
Measure: Mean (Standard Deviation); unit: percentage of correct phonemes
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
Number analyzed (Participants) | 3 | 3
percentage of correct phonemes | 19.75 (28.71) | 16.24 (2.36)
Statistical Analysis 1: Comparison: Stimuli Administered Via 2D Format on an iPad Pro vs Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; Articulation Accuracy does not statistically differ for the iPad Pro or VR goggle participant group after having used the VAST system for 2 months; Test type: Superiority; p = 0.4296, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = -3.51, 95% CI 2-sided [-49.68 to 42.66], Standard Deviation 4.3 — Difference = (VR goggles group - iPad Pro group)
Statistical Analysis 2: Comparison: Stimuli Administered Via 2D Format on an iPad Pro; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.294, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 19.75, 95% CI 2-sided [-25.7 to 65.2], Standard Deviation 24.19 — Difference = (iPad Pro group Post-Treatment - iPad Pro group Pre-Treatment)
Statistical Analysis 3: Comparison: Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.419, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 16.25, 95% CI 2-sided [-33.86 to 66.36], Standard Deviation 19.9 — Difference = (VR goggles group Post-Treatment - VR goggles group Pre-Treatment)

4. Secondary Outcome: Parent Perceptions of Communication Changes, Resulting From Study Participation.
Description: Parent observations -- perceptions of changes in their children's motor-speech, behavioral, and social communication skills after having participated in the study
  Scale title: Net Positive Changes Score Maximum possible value: 18 Minimum possible value: -2 Higher score is better.
Time Frame: as for outcome 1
Population: All participants for each respective group.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Parents of Participants, Who Received VAST Stimuli Via a 2D Format on an iPad Pro: Three parents parents of participants, who received stimuli administered via 2D format on an iPad Pro, answered a 5-question survey, regarding their perceptions of changes in their children's motor-speech, behavioral, and social communication skills after having participated in the study.
- Parents of Participants, Who Received VAST Stimuli Through VR Goggles and Bone Conduction Headphones: Three parents parents of participants -- who received stimuli administered within a 3D format that included VR goggles and bone conduction headphones -- answered a 5-question survey, regarding their perceptions of changes in their children's motor-speech, behavioral, and social communication skills after having participated in the study.
Arm/Group | Parents of Participants, Who Received VAST Stimuli Via a 2D Format on an iPad Pro | Parents of Participants, Who Received VAST Stimuli Through VR Goggles and Bone Conduction Headphones
Number analyzed (Participants) | 3 | 3
Score on a scale | 11 (2.45) | 9.67 (4.18)
Statistical Analysis 1: Comparison: Parents of Participants, Who Received VAST Stimuli Via a 2D Format on an iPad Pro vs Parents of Participants, Who Received VAST Stimuli Through VR Goggles and Bone Conduction Headphones; Test type: Superiority; p < 0.659, ANOVA — Sample size to small for statistical power; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-6.436 to 9.096], Standard Deviation 1.63 — difference = (iPad group mean - VR goggles group mean)

5. Secondary Outcome: Change in Type-Token Ratios
Description: A type-token ratio measures the total number of unique words in a given segment of language.
Time Frame: as for outcome 1
Population: All participants for each respective group.
Measure: Mean (Standard Deviation); unit: number of unique words in a segment
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
Number analyzed (Participants) | 3 | 3
number of unique words in a segment | 30.158 (24.5) | 22.26 (41.18)
Statistical Analysis 1: Comparison: Stimuli Administered Via 2D Format on an iPad Pro vs Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; Test type: Superiority; p < 0.789, ANOVA; Sample size too small for statistical power; Mean Difference (Final Values) = 7.9, 95% CI 2-sided [-68.91 to 84.7], Standard Deviation 9.67 — Difference = (iPad Pro group - VR Goggles group)
Statistical Analysis 2: Comparison: Stimuli Administered Via 2D Format on an iPad Pro; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.304, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 30.16, 95% CI 2-sided [-40.85 to 101.17], Standard Deviation 36.94 — Difference = (iPad Pro group Post-Treatment - iPad Pro group Pre-Treatment)
Statistical Analysis 3: Comparison: Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.403, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 22.26, 95% CI 2-sided [-43.91 to 88.43], Standard Deviation 27.26 — Difference = (VR goggles group Post-Treatment - VR goggles group Pre-Treatment)

6. Secondary Outcome: Increase in Response Rate to Treatment Stimuli
Description: The change in response rate measures any significant differences in how often children responded to pre- and post-testing stimuli after having received treatment between the iPad Pro and VR goggles groups. A response is considered a verbal or non-verbal reaction (e.g., eye contact, gestures, vocalizations) to the stimuli presented during the therapy sessions. Higher response rates indicate better engagement and responsiveness to the treatment. The change in response rate is calculated as the value at the post-test time point minus the value at the pre-test time point, with positive numbers representing increases and negative numbers representing decreases in response rate.
Time Frame: as for outcome 1
Population: All participants for each respective group.
Measure: Mean (Standard Deviation); unit: Number of responses
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
Number analyzed (Participants) | 3 | 3
Number of responses | 5.67 (3.4) | 3.33 (4.03)
Statistical Analysis 1: Comparison: Stimuli Administered Via 2D Format on an iPad Pro vs Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; The response to treatment stimuli will not increase from baseline for the either the iPad Pro or VR goggle participant group after having used the VAST system for 2 months; Test type: Superiority; p < 0.485, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-10.79 to 6.11], Standard Deviation 2.87 — Difference = (VR goggles group - iPad Pro group)
Statistical Analysis 2: Comparison: Stimuli Administered Via 2D Format on an iPad Pro; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.065, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 5.66, 95% CI 2-sided [-0.569 to 11.9], Standard Deviation 6.94 — Difference = (iPad Pro group Post-Treatment - iPad Pro group Pre-Treatment)
Statistical Analysis 3: Comparison: Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones; Comparison of pre-test and post-test outcome per group; Test type: Superiority; p < 0.549, ANOVA — Sample size is too small for statistical power; Mean Difference (Final Values) = 3.34, 95% CI 2-sided [-10.85 to 17.53], Standard Deviation 4.09 — Difference = (VR goggles group Post-Treatment - VR goggles group Pre-Treatment)

ADVERSE EVENTS:
Time Frame: 7 weeks -- each subject participated in the study twice a week over a 7-week period for a total of 14 sessions. The first and last sessions (session #1 and session #14) were reserved for pre-test and post-test language sample collection and assessment.
Description: Our study used a teletherapy platform, which posed no serious risk of physical harm, little to no exposure to psychological harm, social-economic risk, loss of confidentiality, or legal risk.
Arm/Group | Stimuli Administered Via 2D Format on an iPad Pro | Stimuli Administered in 3D Format Via VR Goggles and Bone Conduction Headphones
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
The original research plan called for testing 30 children; however, the pandemic and lockdowns required heavy modification to the research plan. We modified the design to allow subjects to participate in the study remotely. We faced further challenges in recruiting a large enough subject pool, which resulted in our recruiting 10 participants. However, despite our best efforts, the study suffered attrition of four subjects shortly before the beginning, resulting in a final N of 6.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT04764539/Prot_SAP_000.pdf